CLINICAL TRIAL: NCT05600010
Title: Detection of Microplastics in Cardiac Surgery Patients: Its Metabolic Pathways and Toxic Effects
Brief Title: Detection of Microplastics in Cardiac Surgery Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kun Hua (Other)
Responsible Party: Sponsor-Investigator, Kun Hua, Deputy Chief Surgeon, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Other Study IDs: default
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Cardiac Surgery; Microplastics; Nanoplastics; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Microplastics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood; cardiac tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Detection of microplastics/nanoplastics in heart tissue and the blood of patients undergoing cardiac surgery
  Interventions: Other: Microplastics

INTERVENTIONS:
Other: Microplastics — Detection of microplastics as a yes/no value

SUMMARY:
The exponential growth in plastic production/use translates into a parallel increase in environmental plastic waste, which is constantly degraded into microplastics and nanoplastics. Information on the effects of microplastics on human health is still preliminary.

Cardiac surgery patients is a population high exposed to plastics. This observational study will obtain biological samples of cardiac surgery patients as a reference and vulnerable group of individuals highly exposed to microplastics and potentially more susceptible.

The objective of this research is to be able to detect microplastics on blood and operation samples of cardiac surgery patients as well as their potential genotoxic and immunological damage.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Elective cardiac surgery

Exclusion Criteria:

* Emergency surgery or limited-term surgery
* Previous cardiac surgery
* Previous severe liver disease
* Pregnant or planning to become pregnant
* Have a malignant tumor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-10-22 (Estimated)

PRIMARY OUTCOMES:
Detection of microplastics in human heart tissue and the blood | perioperative: preoperative and pro-/postoperative blood and intraoperative heart tissue
  Detection of microplastics in human heart tissue and the blood undergoing cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kun Hua, Study Chair — Beijing Anzhen Hospital